CLINICAL TRIAL: NCT03620708
Title: Addressing Tobacco Use Among Those At Socioeconomic Disadvantage
Brief Title: Tobacco and Socioeconomic Disadvantage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Marc L. Steinberg, Ph.D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro20170000679
Record Dates: First submitted 2018-06-29; First posted 2018-08-08 (Actual); Results first posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Tobacco Smoking
Keywords: tobacco; smoking; cigarette
MeSH Terms: conditions — Tobacco Smoking; Smoking | interventions — Motivational Interviewing; Nicotine Replacement Therapy; Referral and Consultation

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial in which participants are randomized to one of three groups.
Who Masked: Outcomes Assessor
Masking Description: The individual conducting the outcomes assessment is blind to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Motivational Interviewing (Experimental): 35 minute individual motivational interviewing intervention concluding with a written referral sheet for a local smoking cessation clinic and the New Jersey State Quit Line
  Interventions: Behavioral: Motivational Interviewing
- Nicotine Replacement Therapy Sampling (Active Comparator): Participants are provided with a 2-week supply of nicotine patches and a 2 week supply of nicotine lozenges with a recommendation to try them and are also given a written referral sheet for a local smoking cessation clinic and the New Jersey State Quit Line.
  Interventions: Drug: Nicotine Replacement Therapy Sampling
- Referral Only (Other): Participants are provided with a written referral sheet for a local smoking cessation clinic and the New Jersey State Quit Line.
  Interventions: Behavioral: Referral Only

INTERVENTIONS:
Behavioral: Motivational Interviewing — Participants are provided with a 35 minute counseling session designed to increase motivation to quit smoking and then provided with a written referral for tobacco dependence treatment.
  Arms: Motivational Interviewing
Drug: Nicotine Replacement Therapy Sampling — Participants are provided with a two-week sample of over-the-counter nicotine replacement therapy (i.e., nicotine lozenge and nicotine patch) and then provided with a written referral for tobacco dependence treatment.
  Other Names: Nicotine Replacement Therapy
  Arms: Nicotine Replacement Therapy Sampling
Behavioral: Referral Only — Participants are provided with a written referral for tobacco dependence treatment.
  Other Names: Referral
  Arms: Referral Only

SUMMARY:
Randomized clinical trial comparing 3 brief interventions designed to increase motivation to quit smoking in socioeconomically disadvantaged smokers.

DETAILED DESCRIPTION:
The investigators propose a randomized clinical trial comparing 3 brief interventions designed to increase motivation to quit smoking in socioeconomically disadvantaged smokers. Participants will be randomly assigned to receive a) A brief motivational interviewing intervention, b) A nicotine replacement therapy sampling intervention, or c) A referral-only intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the age of 19 and 65
* Participants must self-report being a daily smoker and provide biochemical verification of smoking status (expired breath carbon monoxide reading >5)
* Participants must be at socioeconomic disadvantage, defined as receiving services at a New Brunswick, New Jersey based social services agency (i.e., living in New Brunswick Housing Authority-run public housing units or requesting social services from the community social service agency, "Elijah's Promise")
* Participants must be able to speak and read English.

Exclusion Criteria:

* Participants may not be taking FDA approved smoking cessation or anti-psychotic medications
* Participants may not reported medical issues of potential concern to nicotine replacement users (e.g., unstable angina pectoris, myocardial infarction, or significant cardiac arrythmia (including atrial fibrillation) in the past 30 days)
* Participants may not report pending legal issues with potential to result in incarceration.
* Participants may not be pregnant or nursing, planning on becoming pregnant in the next two months, and must be using effective birth control.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc L Steinberg, Ph.D., Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Division of Addiction Psychiatry, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Motivational Interviewing | Nicotine Replacement Therapy Sampling | Referral Only
Started | 19 | 19 | 20
Completed | 18 | 18 | 17
Not Completed | 1 | 1 | 3
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing | Nicotine Replacement Therapy Sampling | Referral Only | Total
Number analyzed (Participants) | 19 | 19 | 20 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.32 (12.37) | 50.53 (7.97) | 45.65 (10.87) | 47.47 (10.61)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 11 | 14 | 14 | 39
  Female | 7 | 4 | 6 | 17
  Transgender Woman | 1 | 1 | 0 | 2
  Transgender Man | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White / Latinx | 0 | 3 | 3 | 6
  White / Non-Latinx | 10 | 4 | 8 | 22
  Black / Latinx | 0 | 2 | 0 | 2
  Black / Non-Latinx | 7 | 8 | 7 | 22
  American Indian / Alaskan Native and Latinx | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Don't Know / Refused | 2 | 1 | 1 | 4
  Other | 0 | 0 | 1 | 1
  American Indian / Alaskan Native and Not Latinx | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 20 | 58
Cigarettes Per day [Mean (Standard Deviation); unit: cigarettes per day] | 15.47 (6.57) | 11.84 (10.94) | 13.45 (6.58) | 13.59 (8.25)

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Serious Quit Attempt Measured Via the 'Quitting Preparation and Actions Questionnaire'
Description: A self-described "serious" attempt to quit smoking cigarettes since the initial study appointment, measured by the "Quitting Preparation and Actions Questionnaire."
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing | Nicotine Replacement Therapy Sampling | Referral Only
Number analyzed (Participants) | 18 | 18 | 17
Participants | 5 | 10 | 6
Statistical Analysis 1: Comparison: Motivational Interviewing vs Nicotine Replacement Therapy Sampling vs Referral Only; Test type: Superiority; p < 0.05, Chi-squared; chi-square = 3.492

2. Primary Outcome: Self-reported Treatment Seeking Measured Via the 'Quitting Preparation and Actions Questionnaire'
Description: Self-reported contact with one of two treatment referrals provided at intervention since the time of the initial study appointment
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing | Nicotine Replacement Therapy Sampling | Referral Only
Number analyzed (Participants) | 18 | 18 | 17
Participants | 0 | 1 | 3
Statistical Analysis 1: Comparison: Motivational Interviewing vs Nicotine Replacement Therapy Sampling vs Referral Only; Test type: Superiority; p = .113, Chi-squared; chi-square = 4.360

3. Secondary Outcome: Self-reported Cigarettes Per Day
Description: Self-reported cigarettes smoked per day; abstinence to be biochemically verified with carbon monoxide < 5ppm
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: cigarettes/day
Arm/Group | Motivational Interviewing | Nicotine Replacement Therapy Sampling | Referral Only
Number analyzed (Participants) | 18 | 18 | 17
cigarettes/day | 13.0 (7.1) | 7.6 (6.3) | 10.3 (6.9)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Nicotine Replacement Therapy Sampling vs Referral Only; Test type: Superiority; p = .032, ANOVA; Mean Difference (Final Values) = 3.661

4. Secondary Outcome: Importance, Confidence, & Readiness Questionnaire
Description: Motivation and Self-efficacy for quitting smoking measured via Importance, Confidence, & Readiness Questionnaire" (rated on a 0 to 10 scale with higher numbers indicating greater importance, confidence, or readiness to quit)
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Interviewing | Nicotine Replacement Therapy Sampling | Referral Only
Number analyzed (Participants) | 18 | 18 | 17
score on a scale
  Confidence in ability to quit (0-10) | 4.8 (2.8) | 5.5 (3.2) | 6.5 (2.8)
  Importance of Quitting (0-10) | 7.6 (2.9) | 7.3 (3.4) | 8.1 (3.0)
  Readiness to Quit (0-10) | 3.8 (3.1) | 5.1 (3.2) | 5.6 (3.0)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Nicotine Replacement Therapy Sampling vs Referral Only; Examination of differences between groups at follow-up on a measure of confidence in ability to quit; Test type: Superiority; p = .227, ANOVA; Mean Difference (Final Values) = 1.543
Statistical Analysis 2: Comparison: Motivational Interviewing vs Nicotine Replacement Therapy Sampling vs Referral Only; Examination of differences between groups at follow-up on a measure of self-reported importance of quitting smoking; Test type: Superiority; p = .715, ANOVA; Mean Difference (Final Values) = 0.338
Statistical Analysis 3: Comparison: Motivational Interviewing vs Nicotine Replacement Therapy Sampling vs Referral Only; Examination of differences between groups at follow-up on a measure of self-reported readiness to quit smoking; Test type: Superiority; p = .190, ANOVA; Mean Difference (Final Values) = 1.712

5. Secondary Outcome: Readiness to Quit Ladder
Description: "Readiness to Quit Ladder" (with 10 non-numbered choices, ranging from 0 to 10 reflecting varying degrees of readiness to quit smoking; higher numbers reflect greater readiness to quit smoking)
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Motivational Interviewing | Nicotine Replacement Therapy Sampling | Referral Only
Number analyzed (Participants) | 18 | 18 | 17
score on a scale | 5.7 (1.3) | 6.6 (2.1) | 6.4 (2.0)
Statistical Analysis 1: Comparison: Motivational Interviewing vs Nicotine Replacement Therapy Sampling vs Referral Only; Test type: Superiority; p = .188, ANOVA; Mean Difference (Final Values) = 1.728

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Motivational Interviewing | Nicotine Replacement Therapy Sampling | Referral Only
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT03620708/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT03620708/SAP_001.pdf